CLINICAL TRIAL: NCT05794269
Title: Validation of the Turkish Version of QoR-15 (QoR-15T) Scale for Emergency Laparotomy
Brief Title: Turkish Version of the QoR-15 for Emergency Laparotomy
Acronym: QoR-15T-EL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Umut Kara, Associate Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: 2023-20
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life; Anesthesia; Surgery; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Group: Each patient complete the Turkish version of the QoR-15 score (TQoR-15) at 3 times (before surgery, on Day 1, on Day 3).
  Interventions: Other: TQoR-15 questionnaire

INTERVENTIONS:
Other: TQoR-15 questionnaire — The TQoR-15 questionnaire (Turkish version) consists of 15 questions concerning five domains (the patient's feelings, comfort, pain, dependence on the health care team and psychological well-being). Two to three minutes are required to complete all the questions. If the patient is not able to read the questionnaire himself, a third person can ask the patient the questions orally. Each item is scored from 0 to 10 and the total score is the sum of the score obtained for each item, i.e. a score from 0 to 150.

SUMMARY:
Patient perceived quality of recovery is an important outcome after surgery and should be measured in clinical trials. The QoR-15 was designed to measure quality of recovery postoperatively. It provided an efficient evaluation of the postoperative quality of recovery. The primary objectives of this study is validate the Turkish version of QoR-15 questionnaire for emergency laparotomy. The investigators will test its validity, reliability, responsiveness, and clinical acceptability and feasibility, with patients emergency laparotomy, in the University of Health Sciences, Gülhane Education and Training Hospital Ankara, Türkiye.

DETAILED DESCRIPTION:
Recovery from surgery is a complex process that can vary depending on the patient and the anesthesia used. Most clinical studies are interested in reducing perioperative morbidity and mortality, but few evaluate the overall recovery process. The QoR-15 questionnaire assess recovery after elective surgery. A Turkish translation of the QoR-15 score has been validated for use in scheduled surgery. This scale, regardless of the language in which it is translated, has been developed and validated in patients who have undergone scheduled surgery. Until now, no validated scoring tool has been available to assess recovery after emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old,
* Turkish speaking,
* Admitted for any type of emergency laparotomy (time to surgery < 72 hours)
* Able to answer the questionnaire at hospital admission, alone or with the help of a third party
* And agreeing to participate in the study.

Exclusion Criteria:

* Patients with psychiatric or neurological pathologies that compromise cooperation with the protocol,
* Patients admitted for revision surgery,
* aged < 18 years old
* not agreed to provide written informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted for emergency laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Validity of TQoR-15 questionnaire (24 hours) | At 24 hours after surgery
  Evaluate the validity of the Turkish version of the QoR-15 to assess immediate postoperative recovery after emergency laparotomy (at 24 hours)
Validity of TQoR-15 questionnaire (72 hours) | At 72 hours after surgery
  Evaluate the validity of the Turkish version of the QoR-15 to assess immediate postoperative recovery after emergency laparotomy (at 72 hours)

SECONDARY OUTCOMES:
Minimal important difference | At 24 and 72 hours after surgery
  Estimate minimal important difference from the TQoR-15 questionnaire in the emergency laparotomy population.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Gülhane Education and Training Hospital, Etlik, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Kara U, Simsek F, Kamburoglu H, Ozhan MO, Alakus U, Ince ME, Eksert S, Ozkan G, Eskin MB, Senkal S. Linguistic validation of a widely used recovery score: quality of recovery-15 (QoR-15). Turk J Med Sci. 2022 Apr;52(2):427-435. doi: 10.55730/1300-0144.5330. Epub 2022 Apr 14. PMID 36161615